CLINICAL TRIAL: NCT06841016
Title: An Interactive, Conversational Virtual Healthcare Agent to Educate and Engage Patients With Advanced Chronic Kidney Disease About Transplantation (Part 2: Pilot)
Brief Title: Virtual Nephrologist
Acronym: vHCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Florida (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 855462
Record Dates: First submitted 2025-02-10; First posted 2025-02-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease(CKD)
Keywords: CKD; transplantation; virtual healthcare agent; NKF
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Nephrologist (Experimental)
  Interventions: Other: Virtual Nephrologist

INTERVENTIONS:
Other: Virtual Nephrologist — Quality improvement (QI) pilot of an interactive, conversational virtual healthcare agent to educate and engage patients with advanced CKD about transplantation

SUMMARY:
To develop, pilot, and refine a virtual healthcare agent that will educate patients with advanced chronic kidney disease and their caregivers about kidney transplantation.

DETAILED DESCRIPTION:
Over 35 million Americans endure the burdens of chronic kidney disease (CKD). Black Americans face particularly high rates of CKD due to environmental and genetic factors, including systemic racism and inadequate access to specialty providers and effective therapies. The optimal management of advanced CKD poses many challenges for patients, especially those with low health literacy, because of the complexity of medical management and treatment options. For many patients with advanced CKD, pursuing kidney transplantation has major advantages. Compared to chronic dialysis, kidney transplantation improves quality of life and length of life, and offers greater capacity to participate in important activities such as employment. Unfortunately, many patients do not gain sufficient information about kidney transplant or have misconceptions and fears about transplant. This knowledge gap exists in part because many patients have limited access to nephrology care and due to time constraints and ineffective education during nephrology visits. New media technologies can address this need by enabling patients to interact with a virtual health care assistant that both empowers patients to direct the communication toward their own information needs and communicates with patients using language and norms that are comfortable. The study team will develop a virtual healthcare assistant to interact with, educate and counsel patients and their caregivers about kidney transplantation. The tool will provide content developed by the National Kidney Foundation, the leading patient-facing organization focused on kidney disease. Informed by patient partnerships, the tool will address in particular the needs and concerns of Black Americans with kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* 18 y/o able to provide consent
* Advanced CKD
* English speaking
* Penn Medicine patient

Exclusion Criteria:

* Vulnerable populations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Median change in Transplant intention Likert scale question from pre- to post-vHCA | 1 year
  Assess the change in intentionally to consider/discuss getting a kidney transplant using 5-point Likert scale survey

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No